CLINICAL TRIAL: NCT05147025
Title: Evaluation of Retreatment of Failed Revasculatized Teeth by Revascularization. Randomized Clinical Trial
Brief Title: Evaluation of Retreatment of Failed Revasculatized Teeth by Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Principle investigator, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 801
Record Dates: First submitted 2021-10-28; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Revascularization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Revasularization (Experimental): Revascularization of failed previously revascularized younge permenant inciors
  Interventions: Other: Revascularization

INTERVENTIONS:
Other: Revascularization — Regain pulp vascularity for young permenant teeth

SUMMARY:
Study will include 30 participants with failed revascularized young permenant teeth that will be retreated by revascularization and evaluated for success through 2 years

ELIGIBILITY:
Inclusion Criteria:

* central and lateral immature incisors
* child from 8- 10 years old
* healthy chidren
* failed revascularization

Exclusion Criteria:

* medically compromised children
* mentally compromised children

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Root completion | 2 years
  Continue root maturation by radiographic assessment according to cvek classification ( increase root length)
Increase dentine thickness | 2 years
  Increase dentine thickness as response to new formed pulp like tissues
Lesion healing | 2 years
  Resolvation of periapical lesion through new bone formation, intact lamina dura, abscence of periapical radiolucency